CLINICAL TRIAL: NCT05771558
Title: Non-motor Features of Parkinson's Disease
Brief Title: The Effect of a Lighting Intervention on Sleep in Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Rachel Saunders-Pullman, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-22-00991
Record Dates: First submitted 2023-02-21; First posted 2023-03-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease; Sleep Disturbance
MeSH Terms: conditions — Parkinson Disease; Parasomnias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tailored Lighting Intervention (TLI) (Experimental): The TLI will be performed for 2 hours each day over an 8-week period
  During the last week of the lighting, participants will be asked to wear the actigraph and light meter again for 7 days
  Interventions: Device: Tailored Lighting Intervention (TLI); Device: Actigraph

INTERVENTIONS:
Device: Tailored Lighting Intervention (TLI) — The lighting intervention will provide high circadian stimulation produced by light sources that provide moderate light levels of spectra that are tuned to the sensitivity of the circadian system.
Device: Actigraph — An actigraph is a wrist worn devices that measures rest and activity.

SUMMARY:
50 participants with Parkinson's disease will be recruited to complete actigraphy studies to assess sleep disturbances. For this, participants will wear an Actigraph for seven days. Thirty of these participants with sleep disturbance will go on to receive a tailored lighting intervention (TLI) to assess the effect on sleep, fatigue, and circadian entrainment via urinary melatonin levels.

DETAILED DESCRIPTION:
Participants will undergo one week of baseline data collection using the actigraph and light meter and one night of an overnight urine collection. At the completion of the baseline week, the lighting intervention will be installed in the participants' home. Participants will be exposed to the lighting intervention for 2 hours each morning after awakening for 8 weeks. During the last week of the lighting, participants will be asked to wear the actigraph and light meter again for 7 days and collect one overnight urine sample. Participants will complete questionnaires before and after the intervention to further assess its effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease and difficulties with sleep and/or cognition

Exclusion Criteria:

* There are no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Sleep duration using Actigraph | at Baseline for 7 days
  Sleep duration will be calculated by the Actigraph software. A longer sleep duration would indicate an improvement.
Sleep duration using Actigraph | at Week 8 for 7 days
  Sleep duration will be calculated by the Actigraph software. A longer sleep duration would indicate an improvement.

SECONDARY OUTCOMES:
Sleep efficiency using Actigraph | at Baseline for 7 days
  Sleep efficiency will be calculated by the Actigraph software. Sleep efficiency refers to the percentage of time a person sleeps, in relation to the amount of time a spent in bed. The percentage is calculated by dividing actual sleep time by time in bed. A higher sleep efficiency would indicate an improvement.
Sleep efficiency using Actigraph | at Week 8 for 7 days
  Sleep efficiency will be calculated by the Actigraph software. Sleep efficiency refers to the percentage of time a person sleeps, in relation to the amount of time a spent in bed. The percentage is calculated by dividing actual sleep time by time in bed. A higher sleep efficiency would indicate an improvement.
Urine melatonin levels | at Baseline
  Melatonin levels will be assessed from overnight urine collection
Urine melatonin levels | at Week 8
  Melatonin levels will be assessed from overnight urine collection

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Saunders-Pullman, Principal Investigator — Mount Sinai Beth Israel
Locations (1):
- Mount Sinai Beth Israel, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Aggregate results will be published and shared upon request.

DOCUMENTS (1):
  • Informed Consent Form (2024-07-23): https://cdn.clinicaltrials.gov/large-docs/58/NCT05771558/ICF_000.pdf